CLINICAL TRIAL: NCT01350063
Title: Health Impact of Treating and Safely Storing Shallow Tubewell Drinking Water
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR-10038
Record Dates: First submitted 2011-05-04; First posted 2011-05-09 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2011-05

CONDITIONS: Diarrhoeal Disease
Keywords: water; tubewell; diarrhea; chlorination; safe storage
MeSH Terms: conditions — Diarrhea | interventions — troclosene; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Aquatabs and Safe Storage Vessel (Experimental): Households in this group will receive Aquatabs for water purification, a safe water storage container to prevent contamination during storage in the home, and training and encouragement to treat and safely store their water using the provided products.
  Interventions: Drug: Sodium dichloroisocyanurate (NaDCC) tablet (Aquatab)
- Safe Storage Vessel (Experimental): Households in this group will receive a safe water storage container, and training and encouragement to safely store their water using the provided products. If our study shows that treatment of tubewell water at the household level is effective in protecting children's health, they will receive a six-month supply of water treatment tablets at the end of the study.
  Interventions: Device: Water storage container (Jerry can)
- Standard practice (Other): Households in this group will not receive any water treatment or storage intervention during the study. They will continue their usual water collection and storage practices. If our study shows that treatment and safe storage of tubewell water at the household level is effective in protecting children's health, they will receive the same safe water storage container as Groups 1 and 2 as well as a six-month supply of water treatment tablets at the end of the study.
  Interventions: Other: No intervention

INTERVENTIONS:
Drug: Sodium dichloroisocyanurate (NaDCC) tablet (Aquatab) — One tablet should be added to 10L container, resulting in a free chlorine dose of 2 mg/L.
  Other Names: Aquatab
  Arms: Aquatabs and Safe Storage Vessel
Device: Water storage container (Jerry can) — Shallow tubewell water should be stored in 10L container.
  Other Names: Jerry can
  Arms: Safe Storage Vessel
Other: No intervention
  Arms: Standard practice

SUMMARY:
When shallow tubewells replaced highly contaminated surface water as the primary source of drinking water in Bangladesh in the late 20th century, contemporary studies demonstrated no reduction in diarrheal disease with this improvement in water source. This lack of improvement in transitioning to tubewells is consistent with the lack of significant health gains observed in intervention studies focusing on water quality improvements at the source. In contrast, high quality intervention studies that improve water quality at the point of use through treatment of water in households show a 39% reduction in diarrhea.

The primary objective of this study is within a typical setting in rural Bangladesh where households use shallow tubewell water for drinking. The investigators will randomly assign 1800 households who have a child between the ages of six months and two years to one of three groups. Group 1 will receive a safe water storage vessel with a lid and a narrow mouth/tap and Aquatabs, an effervescent water purification tablet that utilizes sodium dichloroisocyanurate (NaDCC) as the chlorine donor. Group 2 will only receive a safe water storage vessel with a lid and a narrow mouth/tap. Group 3 will receive no water intervention and continue their standard habits and practices. Every month a field research assistant will visit each participating household and collect information on the prevalence of diarrhea among children between the ages of six months and two years, as well as children between the ages of two and five years if present in the household. Diarrhea prevalence in the 48 hours and 7 days preceding the visit will be recorded. The investigators will compare the longitudinal prevalence of diarrhea between the following groups: (1) households that receive chlorine and storage container versus households that only receive storage container to assess the effect of chlorination, (2) households that only receive storage container versus households that receive no intervention to assess the effect of safe storage, and (3) households that receive chlorine and storage container versus households that receive no intervention to assess the combined effect of chlorination and safe storage.

Hypothesis:

Drinking water from shallow tubewells that are intermittently contaminated with enteric pathogens contributes importantly to diarrhea among children in rural Bangladesh.

DETAILED DESCRIPTION:
Setting: The investigators will conduct the study in the Fulbaria upazila of Mymensingh district, where groundwater chemistry has been proven to be amenable to disinfection with chlorine. Groundwater in many areas in Bangladesh is rich in iron and other ions that react with chlorine and limit its capacity to provide adequate disinfection. Groundwater testing in Fulbaria has shown that chlorination works effectively at this location, as discussed below.

Develop Intervention: This is an efficacy study, i.e. it is trying to answer the question: if tubewell water were effectively chlorinated and/or safely stored in homes, what would be the impact on childhood diarrhea. To efficiently answer this question, the investigators will strive to optimize the use of the intervention in those households randomized to receive the intervention. Chlorinating water has been shown to be an effective way of disinfecting water in the home (Arnold and Colford, 2007). The investigators will use Aquatabs for chlorination, which are effervescent water purification tablets that utilize sodium dichloroisocyanurate (NaDCC) as the chlorine donor. NaDCC was judged to be a safe and appropriate treatment for water by the World Health Organization (Clasen and Edmondson, 2006) and has been tested and found acceptable to a community of urban residents in Dhaka, Bangladesh (Clasen et al., 2007a). Aquatabs are also easier to store, handle and correctly dose than liquid forms of chlorine (Clasen and Edmondson, 2006).

Groundwater Testing: To optimize the use of Aquatabs and determine the appropriate dose to be assigned to study participants, the investigators collected water samples from 52 shallow tubewells geographically spread out over all 13 unions in Fulbaria. Water was collected in 5L and 10L jerry cans with a narrow mouth and lid. One Aquatabs tablet was added to each vessel, resulting in a free chlorine dose of 2 mg/L in the 10L container and 4 mg/L in the 5L container. Remaining chlorine residual in the vessels was measured half an hour and 24 hours after the addition of the tablet to assess whether it meets the target criteria of having a minimum residual of 0.2 mg/L at 24 hours (to ensure adequate disinfection) and a maximum residual of 2 mg/L at half an hour (to minimize taste and odor concerns). It should be noted that the 2 mg/L taste/odor threshold the investigators are targeting is well under the WHO health limit of 5 mg/L. Based on the testing results, the investigators determined that using one Aquatabs with a 10L jerry can provides the optimal chlorine dose in Fulbaria.

Intervention Groups: The study will have the following three arms, which will allow us to establish the respective roles of household water treatment and safe water storage in preventing diarrheal illness in children in the rural Bangladesh setting.

Group 1 - Aquatabs and Safe Storage Vessel: Households in this group will receive Aquatabs for water purification, a safe water storage container to prevent contamination during storage in the home, and training and encouragement to treat and safely store their water using the provided products.

Group 2 - Safe Storage Vessel: Households in this group will receive a safe water storage container, and training and encouragement to safely store their water using the provided products. If our study shows that treatment of tubewell water at the household level is effective in protecting children's health, they will receive a six-month supply of water treatment tablets at the end of the study.

Group 3 - Standard Practices: Households in this group will not receive any water treatment or storage intervention during the study. They will continue their usual water collection and storage practices. If our study shows that treatment and safe storage of tubewell water at the household level is effective in protecting children's health, they will receive the same safe water storage container as Groups 1 and 2 as well as a six-month supply of water treatment tablets at the end of the study.

Selection of Households: Households to participate in the study will be recruited through a systematic sample from a subset of villages in Fulbaria selected based on field factors such as ease of transport and proximity to the field office. The inclusion criteria will include (1) using a shallow tubewell that is free from iron complaints as the bari's primary source of drinking water and (2) having a child between the ages of six months and two years living in the bari. The primary caregiver in the household that has the child in the target range will be recruited into the study. If there are multiple households in the bari that have a child between the ages of six months and two years, one of the households will be randomly selected and the primary caregiver in the selected household will be recruited. Recruited households will be randomized into one of the three study arms by block randomization through a randomly generated, pre-established sequence that will determine which intervention will be allocated to the household.

Promotion of Interventions: The intervention will continue for five months. At the first visit to the households, Groups 1 and 2 will be provided with a plastic water storage container with a lid and a narrow mouth/tap, and Group 1 will also be given a one-month supply of tablets. Households will be taught through demonstrations and a flipchart with illustrations how to use the tablets as well as how to properly use and clean the safe storage containers, and they will be encouraged to use them regularly. They will also be given an instructions sheet with illustrations that will be left at a visible spot in the household and serve as a reminder to clean the containers and if applicable add the water treatment tablets. A field research assistant who is not part of the evaluation team will visit the household once per month to encourage regular water treatment and safe storage, replenish the supply of tablets and address any issues with the maintenance and cleaning of the safe storage vessels. The rest of the protocol has been written assuming that households will receive monthly promotion visits. However, if the pilot study shows that more frequent, intensive promotion leads to significantly better uptake, in the full-scale study the investigators will consider replacing the monthly promotion frequency with more frequent promotion visits.

Data Collection: There will be one baseline visit and five follow-up visits to participating households.

Baseline Visit: The investigators will conduct a baseline survey including demographics, household description, socioeconomic status, pre-intervention water, sanitation and hygiene habits and baseline levels of diarrhea in children between the ages of six months and two years. If there are any children in a recruited household that are between the ages of two and five, the investigators will collect diarrhea data on them as well to allow comparison of our results to other findings in the literature that focus on children under the age of five. During the baseline visit, the investigators will assess the microbial quality of the tubewell and stored water for each study household using the hydrogen sulphide (H2S) test. Tubewell and stored water samples from a subset of 150 households (50 from each study arm) will be analyzed for total coliforms and E. coli using membrane filtration.

Follow-Up Visits: Every month a field research assistant will visit each participating household to conduct a follow-up survey and collect information on the prevalence of diarrhea among children between the ages of six months and five years in the 48 hours as well as 7 days preceding the visit. The investigators are using a 48-hour recall because this typically provides a more valid estimate than longer recall periods which lead to under-reporting of health outcomes (Alam et al., 1989, Ramakrishnan et al., 1999, Feikin et al., 2010). The investigators are also using a 7-day recall because recent findings indicate that while this longer recall period leads to only minimal bias in terms of the accuracy of recall it can result in significant gains of statistical power (Arnold et al., unpublished data). The investigators will visit households once every month, because more frequent visits provide little additional statistical power due to correlation of repeated measures on the same individuals (Schmidt et al., 2007).

At each visit, the investigators will also collect information on user compliance with the interventions by asking about type and timing of water treatment practices, counting the number of remaining tablets and inspecting the water storage facilities, as well as asking participants when and how they cleaned the storage container. The investigators will also collect water samples from the tubewell and storage container in households to assess the microbial quality of the water, explore the extent of contamination at the source versus in the home and gauge the effectiveness of the interventions in preventing contamination. The investigators will perform H2S testing in half of study households and total coliform/E.coli testing with membrane filtration for a subset of 150 households (50 from each study arm). Moreover, for each household in the Aquatabs group, the investigators will analyze stored water samples for residual chlorine concentration to monitor compliance with the intervention.

Laboratory Testing: Water samples will be placed on ice and transported to the Fulbaria field office where the appropriate tests will be conducted by the field microbiologists. All testing will be performed promptly upon transporting the samples to the field office. The hydrogen sulfide (H2S) test is a simple low-cost test (Sobsey and Pfaender, 2003). Twenty ml of water will be added in H2S bottle and incubated at room temperature for 24-48 hours. If the colour of the water changes to black, it will indicate that the water is contaminated with coliform which will indicate that the water is unfit for human consumption. For membrane filtration, collected water samples will be quantitatively tested for total coliforms and E. coli using the DelAgua kit with MI Broth (Whatman Inc, New Jersey, USA). For residual chlorine testing, the investigators will use the n,n-diethyl-p-phenylenediamine (DPD) colorimetric method which is part of the DelAgua kit.

ELIGIBILITY:
Inclusion Criteria:

* Using a shallow tubewell that is free from iron complaints as the bari's primary source of drinking water and
* Having a child between the ages of six months and two years living in the bari

Exclusion Criteria:

* Iron complaints of the shallow tubewell

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1800 (Actual)
Dates: Start 2011-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Diarrhoeal incidence among children between 6 months to 5 years of age. | 6 months
  6 months' intervention. Follow-up will be done once in a month. Information on diarrhoeal episodes will be collected for 7 days prior to the follow-up day.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Luby, MD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Fulbaria sub-district, Mymensingh, Bangladesh

REFERENCES:
- [Derived] Ercumen A, Naser AM, Unicomb L, Arnold BF, Colford JM Jr, Luby SP. Effects of source- versus household contamination of tubewell water on child diarrhea in rural Bangladesh: a randomized controlled trial. PLoS One. 2015 Mar 27;10(3):e0121907. doi: 10.1371/journal.pone.0121907. eCollection 2015. PMID 25816342